CLINICAL TRIAL: NCT04406051
Title: Prevention of Maternal Hypotension During Cesarean Section With Norepinephrine Infusion. Does Time and Type of Administered Fluids Matter?
Brief Title: Prevention of Maternal Hypotension During Cesarean Section With Norepinephrine Infusion.
Acronym: annie-manos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aretaieion University Hospital (Other)
Collaborators: Alexandra Hospital, Athens, Greece (Other)
Responsible Party: Principal Investigator, Dr Kassiani Theodoraki, Professor of Anesthesiology, Aretaieion University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: nor-cryst vs. nor-coll
Record Dates: First submitted 2020-05-24; First posted 2020-05-28 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Hypotension; Obstetric Anesthesia Problems; Cesarean Section Complications; Hypotensive; Vasoconstriction
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- norepinephrine infusion and colloid preloading (NOR-COL) (Active Comparator): in parturients allocated to the NOR-COL group, a norepinephrine infusion will be started as soon as spinal anesthesia is initiated. This group will also receive colloid preloading (5 mL/kg)
  Interventions: Procedure: norepinephrine infusion and colloid preloading (NOR-COL)
- norepinephrine infusion and crystalloid co-loading (NOR-CRYS) (Active Comparator): in parturients allocated to the NOR-CRYST group, a norepinephrine infusion will be started as soon as spinal anesthesia is initiated. This group will also receive crystalloid co-loading (10 mL/kg)
  Interventions: Procedure: norepinephrine infusion and crystalloid co-loading (NOR-CRYST)

INTERVENTIONS:
Procedure: norepinephrine infusion and colloid preloading (NOR-COL) — in parturients allocated to the NOR-COL group, a norepinephrine infusion will be started as soon as spinal anesthesia is initiated. This group will also receive 5 mL/kg of colloid infusion prior to the initiation of spinal anesthesia
  Arms: norepinephrine infusion and colloid preloading (NOR-COL)
Procedure: norepinephrine infusion and crystalloid co-loading (NOR-CRYST) — in parturients allocated to the NOR-CRYST group, a norepinephrine infusion will be started as soon as spinal anesthesia is initiated. This group will also receive 10 mL/kg of crystalloid infusion simultaneously with the initiation of spinal anesthesia
  Arms: norepinephrine infusion and crystalloid co-loading (NOR-CRYS)

SUMMARY:
This will be a randomized study aiming at investigating the combination of a norepinephrine infusion and colloid preloading versus the combination of a norepinephrine infusion and crystalloid co-loading for the prevention of maternal hypotension during elective cesarean section

DETAILED DESCRIPTION:
Neuraxial techniques are the anesthetic techniques of choice in contemporary obstetric anesthesia practice, with a definitive superiority as compared to general anesthesia, since, by their use, serious complications involving the airway can be avoided.Spinal anesthesia has become the favorable technique for both elective and emergency cesarean section due to a quick and predictable onset of action, however, it can be frequently complicated by hypotension, with incidence exceeding 80% occasionally. Recently, noradrenaline has been shown to be effective in maintaining blood pressure in obstetric patients. Another technique widely used to prevent hypotension is fluid administration. Current evidence suggests that the combination of fluid administration and vasoconstrictive medications should be the main strategy for prevention and management of hypotension accompanying neuraxial anesthesia procedures during cesarean section. Research is still underway in relation to the most appropriate timing for fluid administration, the most appropriate fluid volume as well as the type of fluid that should be administered. However, preloading of crystalloids seems to be inefficient as a sole strategy, while co-loading of colloids is more effective than co-loading of crystalloids for prevention of hypotension in the parturient. On the other hand, preloading and co-loading of colloids seem to be of equal effectiveness. Literature is rather scarce regarding the comparison of colloid preloading and crystalloid co-loading.

The aim of this randomized study will be to investigate the combination of a norepinephrine infusion and colloid preloading versus the combination of a norepinephrine infusion and crystalloid co-loading for the prevention of maternal hypotension during elective cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* adult parturients, American Society of Anesthesiologists (ASA) I-II,
* singleton gestation>37 weeks
* elective cesarean section

Exclusion Criteria:

* Body Mass Index (BMI) >40 kg/m2
* Body weight <50 kg
* Body weight>100 kg
* height<150 cm
* height>180 cm
* multiple gestation
* fetal abnormality
* fetal distress
* active labor
* cardiac disease
* pregnancy-induced hypertension
* thrombocytopenia
* coagulation abnormalities
* use of antihypertensive medication during pregnancy
* communication or language barriers
* lack of informed consent
* contraindication for regional anesthesia

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2020-05-26 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
incidence of hypotension | intraoperative
  any occurence of hypotension (systolic blood pressure<80% of baseline) throughout the operation will be recorded

SECONDARY OUTCOMES:
need for vasoconstrictor | intraoperative
  any need for vasoconstrictor during the operation will be recorded
type of vasoconstrictor administered | intraoperative
  phenylephrine versus ephedrine
total dose of vasoconstrictor administered | intraoperative
  total dose in mg for ephedrine or μg for phenylephrine administered
incidence of hypertension | intraoperative
  any incidence of systolic blood pressure>120% of baseline will be recorded
incidence of bradycardia | intraoperative
  any incidence of maternal bradycardia (heart rate<60/min) will be recorded
need for atropine | intraoperative
  any need for atropine during the operation because of bradycardia will be recorded
modification or cessation of the infusion | intraoperative
  any requirement for modification or cessation of the infusion due to reactive hypertension or bradycardia will be recorded
incidence of nausea/vomiting | intraoperative
  any occurence of nausea and/or vomiting during the operation will be recorded
Neonatal Apgar score at 1 min | 1 min post delivery
  Neonatal Apgar score will be recorded at 1 min after delivery. The Apgar score is determined by evaluating the newborn baby on five simple criteria on a scale from zero to two, then summing up the five values thus obtained. The resulting Apgar score ranges from zero to 10. Scores 7 and above are generally normal; 4 to 6, fairly low; and 3 and below are generally regarded as critically low and cause for immediate resuscitative efforts.
Neonatal Apgar score at 5 min | 5 min post delivery
  Neonatal Apgar score will be recorded at 5 min after delivery. The Apgar score is determined by evaluating the newborn baby on five simple criteria on a scale from zero to two, then summing up the five values thus obtained. The resulting Apgar score ranges from zero to 10. Scores 7 and above are generally normal; 4 to 6, fairly low; and 3 and below are generally regarded as critically low and cause for immediate resuscitative efforts.
neonatal blood gases | 1 min post delivery
  fetal cord blood analysis will be performed immediately post-delivery
glucose in neonatal blood | 1 min post delivery
  glucose will be measured in the cord blood gas sample taken immediately post-delivery

CONTACTS AND LOCATIONS:
Overall Officials: Kassiani Theodoraki, PhD, DESA, Principal Investigator — Aretaieion University Hospital; Emmanouil Stamatakis, PhD, Principal Investigator — Alexandra General Hospital of Athens; Sofia Hadzilia, MD, Principal Investigator — Alexandra General Hospital of Athens; Dimitrios Valsamidis, MD, Principal Investigator — Alexandra General Hospital of Athens; Konstantina Kalopita, MD, Principal Investigator — Alexandra General Hospital of Athens
Locations (2):
- Greece (2):
  - Aretaieion University Hospital, Athens
  - Alexandra General Hospital of Athens, Athens

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Afolabi BB, Lesi FE. Regional versus general anaesthesia for caesarean section. Cochrane Database Syst Rev. 2012 Oct 17;10(10):CD004350. doi: 10.1002/14651858.CD004350.pub3. PMID 23076903
- [Background] Klohr S, Roth R, Hofmann T, Rossaint R, Heesen M. Definitions of hypotension after spinal anaesthesia for caesarean section: literature search and application to parturients. Acta Anaesthesiol Scand. 2010 Sep;54(8):909-21. doi: 10.1111/j.1399-6576.2010.02239.x. Epub 2010 Apr 23. PMID 20455872
- [Background] Ngan Kee WD. Prevention of maternal hypotension after regional anaesthesia for caesarean section. Curr Opin Anaesthesiol. 2010 Jun;23(3):304-9. doi: 10.1097/ACO.0b013e328337ffc6. PMID 20173633
- [Background] Kinsella SM, Carvalho B, Dyer RA, Fernando R, McDonnell N, Mercier FJ, Palanisamy A, Sia ATH, Van de Velde M, Vercueil A; Consensus Statement Collaborators. International consensus statement on the management of hypotension with vasopressors during caesarean section under spinal anaesthesia. Anaesthesia. 2018 Jan;73(1):71-92. doi: 10.1111/anae.14080. Epub 2017 Nov 1. No abstract available. PMID 29090733
- [Background] Banerjee A, Stocche RM, Angle P, Halpern SH. Preload or coload for spinal anesthesia for elective Cesarean delivery: a meta-analysis. Can J Anaesth. 2010 Jan;57(1):24-31. doi: 10.1007/s12630-009-9206-7. Epub 2009 Oct 27. PMID 19859776
- [Background] Mercier FJ. Fluid loading for cesarean delivery under spinal anesthesia: have we studied all the options? Anesth Analg. 2011 Oct;113(4):677-80. doi: 10.1213/ANE.0b013e3182245af4. No abstract available. PMID 21948275
- [Background] Li L, Zhang Y, Tan Y, Xu S. Colloid or crystalloid solution on maternal and neonatal hemodynamics for cesarean section: a meta-analysis of randomized controlled trials. J Obstet Gynaecol Res. 2013 May;39(5):932-41. doi: 10.1111/jog.12001. Epub 2013 Feb 4. PMID 23379937